CLINICAL TRIAL: NCT02959541
Title: An Open Randomized Single Site Pharmacokinetic and Pharmacodynamic Study, of Calciumfolinat 60 mg/m², 200 mg/m² or 500 mg/ m² in Blood, Tumor and Adjacent Mucosa From Patients With Colon Cancer
Brief Title: PK/PD Investigation of Calciumfolinat in Blood, Tumor and Adjacent Mucosa in Patient With Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00068128
Record Dates: First submitted 2016-10-20; First posted 2016-11-09 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2021-09

CONDITIONS: Colon Cancer; Chemotherapy
Keywords: Leukovorin
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Calciumfolinat 60 mg/m² (Other): Intravenous infusion of Calciumfolinat 60 mg/m²given to patients with colon cancer at the time for the operation of the colon cancer.
  Interventions: Drug: Leucovorin
- Calciumfolinat 200 mg/m² (Other): Intravenous infusion of Calciumfolinat 200 mg/m² given to patients with colon cancer at the time for the operation of the colon cancer.
  Interventions: Drug: Leucovorin
- Calciumfolinat 500 mg/ m² (Other): Intravenous infusion of Calciumfolinat 500 mg/ m² given to patients with colon cancer at the time for the operation of the colon cancer.
  Interventions: Drug: Leucovorin

INTERVENTIONS:
Drug: Leucovorin
  Other Names: Calciumfolinat is the brandname of Leucovorin

SUMMARY:
This is an open randomized single site Pharmacokinetic and Pharmacodynamic study,of Calciumfolinat 60 mg/m², 200 mg/m² or 500 mg/ m² in blood, tumor and adjacent mucosa from patients with colon cancer

DETAILED DESCRIPTION:
Cytotoxic treatment of patients with colorectal cancer (CRC) includes most various different drugs but 5-fluorouracil (5-FU) is the cornerstone in most regimens. Leucovorin (LV) is frequently used as a part of a standard treatment regime for advanced CRC in combination with 5-FU. In numerous randomized clinical trials the addition of LV to 5-FU has been shown to significantly improve the antitumor activity and to prolong the survival of patients receiving adjuvant chemotherapy or treatment for advanced disease as to compared to treatment with 5-FU as single drug therapy.

In most European countries 5-FU is given as an infusion during 46 hours in combination with a two hour infusion of LV. This regime is called the deGramont schedule. In the Nordic countries, 5-FU and LV are often given as bolus injections according to the regime called Nordic FLV. Leucovorin is a prodrug which has to be metabolized to methylenetetrahydrofolate (mTHF) in order to increase inhibition of the target enzyme thymidylate synthase (TS). Due to the low concentrations of the reduced folate forms intracellular there is a lack of knowledge of the pharmacodynamics of LV when used as an infusion. When the 5-FU/LV used today was introduced it was technically not possible to measure the different metabolites of the reduced folates in blood and tissue. In the literature there is only one published reference measuring the blood concentration after a two hour infusion of LV. However, it has recently been possible to separate and quantitate the different folates using sensitive Liquid Chromatography/Masspectrometry (LC/MS) methods. Furthermore it has been stated that differences in enzyme activity for genes involved in the transport and metabolism of folates may be responsible for the large inter individual differences in folate tissue concentrations.

This study is designed to gain an understanding of how a single intravenous infusion of LV affects the folate concentration in blood, tumor and adjacent mucosa tissue. By using the LC/MS method which was recently developed and it is now possible to quantitate the different metabolites of LV in small tissue samples as well as in blood. It is further now possible to measure by quantitative Polymerase Chain Reaction techniques (PCR) the most important genes involved in the folate transport and metabolism ((SHMT1), SerineHydroxyMethylTransferase1 and (ABCC3) ATP-binding cassette, sub-family C, (CFTR/MRP), member 3)).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an operable colon cancer that is determined to colorectal surgery
2. Patients must sign an informed consent document
3. Patients must be ≥ 18 years of age
4. Fertile women must present a negative pregnancy test and use secure contraceptives during and three months after treatment

Exclusion Criteria:

1. Neo-adjuvant chemotherapy within the last 30 days
2. Presence of clinically relevant (i.e., detectable by physical examination) third-space fluid collection (e.g., ascites, pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry
3. Female patients: currently pregnant or breast-feeding
4. Patient with epileptic medication, such as fenobarbital, primidon, fenytoin och succinimider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
[6R] 5,10-methylene-THF - tumor | First day during surgery
  Tissue concentration of [6R] 5,10-methylene-THF in the tumor
[6R] 5,10-methylene-THF - adjacent mucosa | First day during surgery
  Tissue concentration of [6R] 5,10-methylene-THF in adjacent mucosa
5-formyl-THF - tumor | First day during surgery
  Tissue concentration of 5-formyl-THF in the tumor
5-formyl-THFin - adjacent mucosa | First day during surgery
  Tissue concentration of 5-formyl-THFin the adjacent mucosa
5-methyl-THF - tumor | First day during surgery
  Tissue concentration of 5-methyl-THF in the tumor
5-methyl-THF - adjacent mucosa | First day during surgery
  Tissue concentration of 5-methyl-THF in the adjacent mucosa
THF - tumor | First day during surgery
  Tissue concentration of THF in the tumor
THF - adjacent mucosa | First day during surgery
  Tissue concentration of THF in the adjacent mucosa

SECONDARY OUTCOMES:
AUC [6R] 5,10-methylene-THF | Up to 24 hours
  AUC(0-24h) calculated from plasma concentration of [6R] 5,10-methylene-THF
AUC 5-formyl-THF | Up to 24 hours
  AUC(0-24h) calculated from plasma concentration of 5-formyl-THF (if data
AUC 5-methyl-THF | Up to 24 hours
  AUC(0-24h) calculated from plasma concentration of 5-methyl-THF (if data permits)
AUC THF | Up to 24 hours
  AUC(0-24h) calculated from plasma concentration of THF (if data permits)
Correlation AUC - blood and tissue | Up to 24 hours
  Correlation between AUC calculated from blood concentration and tissue concentration in the tumor and adjacent mucosa
Gene expression - correlation to tissue concentration of the reduced folates | First day during surgery
  Gene expression in the tumor and correlation to tissue concentration of the reduced folates
Gene expression - correlation adjacent mucosa tissue concentration of the reduced folates | First day during surgery
  Gene expression in the adjacent mucosa and correlation to tissue concentration of the reduced folates

CONTACTS AND LOCATIONS:
Overall Officials: Elinor Bexe Lindskog, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of surgery, Östra, Sahlgrenska University Hospital, Gothenburg, Sweden